CLINICAL TRIAL: NCT02163044
Title: A Study to Assess the Consequences of Postprandial Lipemia in CRP as Inflammatory Marker in High-risk Adults, to Investigate Whether Hypolipidemic, Hypoglycemic or Antihypertensive Medication May Lessen the Exaggerated Postprandial Lipemia and Evaluate the Influence of Gene Polymorphisms Involved in Lipid and Glucose Metabolism on Postprandial Lipemia and Cardiovascular Outcomes.
Brief Title: The Hellenic Postprandial Lipemia Study (HPLS)
Acronym: HPLS
Status: Completed | Type: Observational
Sponsor: Hellenic College of Treatment of Atherosclerosis (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-HPLS-IIS
Record Dates: First submitted 2014-06-04; First posted 2014-06-13 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Coronary Heart Disease; Dyslipidemia
MeSH Terms: conditions — Coronary Disease; Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Statin: Patients on statin treatment

SUMMARY:
Coronary heart disease (CHD) is the leading cause of death worldwide. The disease is characterized by a high mortality rate (about 40%) and a course continuously altered by lifestyle, gene polymorphisms and therapeutic treatment. Fasting concentration of blood lipids and lipoproteins only partially express the complex relation between dyslipidemia and CHD. Following the indication stated nearly 40 years ago by Zilversmit, there is now accumulating evidence that postprandial lipemia plays an important role in the atherogenic process [ref Kolovou], particularly that most hours of the day are spent in the postprandial state. Furthermore, the increases in blood glucose and triglycerides (TGs) following meals stimulate oxidative stress, impair endothelial function, and rises the inflammatory factors that lead to atherosclerosis. Previous studies reported on postprandial lipemia in subjects with obesity, metabolic syndrome, diabetes mellitus, elderly, patients with CHD and others. However, currently the estimation of cardiovascular disease risk is based on fasting blood values of triglycerides (TGs) and inflammatory markers. The effect of postprandial atherogenic factors on the initiation and progression of atherosclerosis is actually not known.The Hellenic Postprandial Lipemia Study (HPLS) was designed to study the consequences of postprandial lipemia in CRP as inflammatory marker in high-risk adults. Furthermore, the HPLS study will investigate whether hypolipidemic, hypoglycemic or antihypertensive medication may lessen the exaggerated postprandial lipemia as well as the rest abnormal postprandial metabolism. Finally, the HPLS study is intending to evaluate the influence of gene polymorphisms involved in lipid and glucose metabolism on postprandial lipemia and cardiovascular outcomes.

DETAILED DESCRIPTION:
The study aims to recruit 1200 patients that are characterized either as high risk or very-high risk for Coronary Heart Disease. It is assumed that an equal number of high risk and very high risk patients will be included in the study. Patients will be invited to participate in the study from outpatient clinics in the 14 centers in Athens, Greece.

The study will be approved by the institution ethics committee and informed consent will be obtained from all participating patients.

Participating patients will have recently (up to 15 days) been initiated in one of the following dislipidemic treatments:

* Simvastatin up to 40 mg,
* Atorvastatin up to 80 mg,
* Rosuvastatin up to 40 mg,
* Statin intolerant subjects receiving colesevelam up to 3.75 g/day or fenofibrate 145 mg/day.

All patients should have received the above treatments as initial treatment for dyslipidemia with the exception of statin intolerant patients. All patients at the time of their inclusion in the study will have been evaluated for gene polymorphisms as part of their dyslipidemic profile evaluation. Furthermore patients will have been characterized as high risk or very high risk according to the SCORE level of risk, calculated using the Greek version of low-risk regions charts.

Each center will recruit 50 very high and 50 high risk patients. Each site will include 10 consecutive high risk and 10 very high risk patients for each treatment group as described above. The following data will be collected for each patient:

* Personal and demographic details
* Family and personal medical history (including smoking, hypertension, hyperlipidemia and glucose metabolism, as well as cardiovascular disease history)
* Past measurements of blood pressure,
* Diabetes and lipids,
* Diagnostic procedures undertaken (coronary or other angioplasty, Coronary artery by-pass surgery),
* Measurements of blood pressure,
* Weight, height, waist and hip circumference. Body mass index (BMI) will be calculated as weight/height2
* The SCORE level of risk will be also calculated using the Greek version of low-risk regions charts.

Each subject will have to complete 2 Lipotest meals with the first one given at the beginning of the study and the second one after at least 3 months of hypolipidemic treatment. Before and 4 hours after the meals blood samples will be collected. After that, subjects will be followed annually for 3 years.

Lipotest Meal The Lipotest meal is a diagnostic standardized meal recognized by Hellenic Drug Organization (EOF, National Drug Organization). A single serving, provided in a sachet, is comprised of 115 g powder that is rehydrated by adding 150 ml water.

The powder and water are mixed to homogeneity (2-3 minutes with a hand held mixer), and then refrigerated to form a mousse. All ingredients are food grade and are stable for a period of 24hours after preparation as proved by antioxidant tests The ingredients' composition of Lipotest is hydrogenated vegetable fat, glucose syrup solids, milk proteins, sugar, emulsifiers (lactic and acetic acid esters of monoglycerides and diglycerides, cocoa powder (20-22% fat content), defatted cocoa powder (10-12% fat content), and flavorings.

On a per serving basis, Lipotest provides 832 kcal (42% FDA Daily reference value (DRV) for adults, and 42% of the European Guideline Daily Amount, GDA), 10 g protein (20% DRV, 20% GDA), 25 g of carbohydrates (8.3% DRV, 10% GDA) of which simple sugars comprise 14.3 g (no DRV, 16% GDA), 2.1 g fiber (8.4% DRV), 0.15 g salt (2.5% DRV for sodium), and 75 g fat (115 % DRV, 109% GDA), all of which is fully saturated (375% DRV and GDA) through hydrogenation of vegetable fat. Fat used is coconut oil named Cegepal VF HC 77 and Lamequick 6068 both from Cognis, which are fully approved for use in food applications and are in powder form.

Oral fat loading The meal will be administrated in the morning after 12-h overnight fast. Subjects will eat meal within 20 min and will be instructed to keep physical activity to a minimum, refrain from smoking and fast during the 4 h of the test. Blood samples will be withdrawn at 0 and 4 h for determination of TGs concentration. The meal will be administrated twice, before any treatment (visit 1) and 3 months after treatment with hypolipidemic, hypoglycemic or antihypertensive drugs (visit 2).

Collection of blood and biomarker analyses All laboratory tests will be carried out at as part of everyday clinical practice and will be covered by the patient insurance.

Serum total cholesterol (TC), high density lipoprotein cholesterol (HDL-C) and TG concentrations will be measured from both fasting and postprandial blood samples and plasma glucose concentrations will be measured from true fasting blood samples only.

Inflammatory marker analysis Plasma will be analyzed for hs-C-reactive protein (CRP) according to everyday clinical practice and will be covered by the patient insurance.

Study Duration 18 months recruitment period. 3 years follow up for every patient.

Subject Participation Duration 36 Months 1200 very high and high risk for CHD patients

Number of Participating Sites 14 clinics in 12 Hospitals

Investigational Product: Not Applicable Investigational Product Dosage & Administration: Not Applicable

Concomitant Medication All patients will receive concomitant medication in accordance to the everyday practice of their treating physician.

Safety Evaluation All adverse events will be recorded in accordance to all applicable laws and regulations concerning medications prescribed according to their approved summary of product characteristics.

Statistical Analysis Continuous variables will be described using means and standard deviations. Comparisons of continuous variables will be performed using the Student's t-test or the Mann-Whitney-U test for parametric and non-parametric data, respectively. Categorical variables will be expressed as absolute (N) or relative (%) frequencies and will be analyzed for associations using the chi-square test. The Paired t-test will be used to compare changes within the groups of variables and the Bonferroni test will be used to compare the changes between the groups, as a method for their post hoc comparisons Univariate and multivariate stepwise linear regression analyses will be performed in order to identify independent predictors for CRP and other dependent variables.

Survival analysis will be performed to elucidate potential predictors of MACE using both fasting and postprandial values of the studies variables and gene polymorphisms.

All tests will be two-sided. P-value will be considered statistically significant if <0.05. Data will be analyzed using STATA™ statistical software (Version 9.0, Stata Corporation, College Station, TX 77845, USA).

Ethical Considerations The Ethics Committee of the each participating Hospital will approve the non interventional study. All participants will sign the written informed consent prior to participation in the study. The information protection rules in the National Institute for Health and Welfare (former National Public Health Institute to 2009) will be followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age,
* Signed informed consent form
* Fasting triglycerides (TGs) < 220 mg/dl
* Liver function tests within normal range
* No more than mild renal impairment (clearance of creatinine >60 ml/min)
* features of very high risk
* documented cardiovascular disease by invasive or non-invasive testing (such as coronary angiography, nuclear imaging, stress echocardiography, carotid plaque on ultrasound)
* previous myocardial infarction
* acute coronary syndrome
* coronary revascularization (percutaneous coronary intervention, coronary artery bypass graft) and other arterial revascularization procedures
* ischemic stroke
* peripheral artery disease
* patients with type 2 diabetes
* patients with type 1 diabetes with target organ damage
* calculated 10 year risk SCORE ≥10%] or
* high risk, markedly elevated single risk factors such as:
* familial dyslipidemias and severe hypertension
* calculated SCORE ≥5% and <10%

Exclusion Criteria:

* history of liver, kidney, pancreas, or gall bladder disease,
* history of acute coronary syndrome one month prior to entering the study
* pregnancy
* presence of any inflammatory disease
* treatment with medications known to affect TGs metabolism or concentration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to recruit 1200 patients that are characterized either as high risk or very-high risk for Coronary Heart Disease. It is assumed that an equal number of high risk and very high risk patients will be included in the study. Patients will be invited to participate in the study from outpatient clinics in the 14 centers in Athens, Greece.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in CRP levels | 0,6,12,18,24,30,36 months
  To study the consequences of postprandial lipemia in CRP as inflammatory marker in high-risk adults.
Change in exaggerated postprandial lipemia | 0,3,6,12,18,24,30,36 months
  To investigate whether hypolipidemic, hypoglycemic or antihypertensive medication may lessen the exaggerated postprandial lipemia as well as the rest abnormal postprandial metabolism.
Change in Lipotest meal values | 0,3,6,12,18,24,30,36 months
  To study the impact of postprandial lipemia using a novel test (Lipotest meal) that distinguishes very-high and high risk subjects in to two subgroups according to first Lipotest meal: the positive group with TG postprandial ≥220 mg/dl, and the negative group with TG postprandial < 220 mg/dl (Consensus criteria).

SECONDARY OUTCOMES:
Number of major adverse cardiovascular events | 0-36 months
  To report on major adverse cardiovascular events (MACE: death from cardiovascular causes, non-fatal myocardial infarction and non-fatal stroke) in subjects in the positive and negative group.

OTHER OUTCOMES:
SCORE prediction model value measurement | 0 - 36 months
  To validate a risk prediction model (SCORE) in order to compare the results from the HPLS study with the results expected to be from the SCORE prediction model.

CONTACTS AND LOCATIONS:
Overall Officials: Genovefa Kolovou, M.D., Ph.D., F.E.S.C., S.F.S.A, Study Director — Onassis Cardiac Surgery of Athens
Locations (1):
- Onassion Cardiology Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tunstall-Pedoe H, Kuulasmaa K, Amouyel P, Arveiler D, Rajakangas AM, Pajak A. Myocardial infarction and coronary deaths in the World Health Organization MONICA Project. Registration procedures, event rates, and case-fatality rates in 38 populations from 21 countries in four continents. Circulation. 1994 Jul;90(1):583-612. doi: 10.1161/01.cir.90.1.583. PMID 8026046
- [Background] Zilversmit DB. Atherogenesis: a postprandial phenomenon. Circulation. 1979 Sep;60(3):473-85. doi: 10.1161/01.cir.60.3.473. PMID 222498
- [Background] Kolovou GD, Anagnostopoulou KK, Daskalopoulou SS, Mikhailidis DP, Cokkinos DV. Clinical relevance of postprandial lipaemia. Curr Med Chem. 2005;12(17):1931-45. doi: 10.2174/0929867054546609. PMID 16101498
- [Background] Tentolouris N, Eleftheriadou I, Katsilambros N. The effects of medications used for the management of dyslipidemia on postprandial lipemia. Curr Med Chem. 2009;16(2):203-17. doi: 10.2174/092986709787002763. PMID 19149572
- [Background] Ceriello A. Effects of macronutrient excess and composition on oxidative stress: relevance to diabetes and cardiovascular disease. Curr Atheroscler Rep. 2006 Nov;8(6):472-6. doi: 10.1007/s11883-006-0022-z. PMID 17045073
- [Background] Kolovou GD, Bilianou H, Mikhailidis DP. Postprandial lipemia in children and adolescents. Curr Vasc Pharmacol. 2011 May;9(3):318-20. doi: 10.2174/157016111795495521. PMID 21314624
- [Background] Burdge GC, Calder PC. Plasma cytokine response during the postprandial period: a potential causal process in vascular disease? Br J Nutr. 2005 Jan;93(1):3-9. doi: 10.1079/bjn20041282. PMID 15705218
- [Background] Ceriello A, Quagliaro L, Piconi L, Assaloni R, Da Ros R, Maier A, Esposito K, Giugliano D. Effect of postprandial hypertriglyceridemia and hyperglycemia on circulating adhesion molecules and oxidative stress generation and the possible role of simvastatin treatment. Diabetes. 2004 Mar;53(3):701-10. doi: 10.2337/diabetes.53.3.701. PMID 14988255
- [Background] Bansal S, Buring JE, Rifai N, Mora S, Sacks FM, Ridker PM. Fasting compared with nonfasting triglycerides and risk of cardiovascular events in women. JAMA. 2007 Jul 18;298(3):309-16. doi: 10.1001/jama.298.3.309. PMID 17635891
- [Background] Kolovou GD, Mikhailidis DP, Kovar J, Lairon D, Nordestgaard BG, Ooi TC, Perez-Martinez P, Bilianou H, Anagnostopoulou K, Panotopoulos G. Assessment and clinical relevance of non-fasting and postprandial triglycerides: an expert panel statement. Curr Vasc Pharmacol. 2011 May;9(3):258-70. doi: 10.2174/157016111795495549. PMID 21314632
- [Derived] Kolovou G, Giannakopoulou V, Kalogeropoulos P, Anagnostopoulou K, Goumas G, Kazianis G, Limberi S, Perrea D, Mihas C, Kolovou V, Bilianou H. Hellenic Postprandial Lipemia Study (HPLS): Rationale and design of a prospective, open-label trial to determinate the prevalence of abnormal postprandial lipemia as well as its interaction with statins in patients at high- and very high-risk for cardiovascular disease. Contemp Clin Trials. 2019 Jul;82:101-105. doi: 10.1016/j.cct.2019.05.011. Epub 2019 May 29. PMID 31150799